CLINICAL TRIAL: NCT04902365
Title: Neurofeedback for Patients With Visual Snow
Brief Title: Neurofeedback in Visual Snow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NeurofeebackSnow
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Visual Snow Syndrome; Neuro-Ophthalmology
Keywords: neurofeedback; real-time functional magnetic resonance imaging
MeSH Terms: conditions — visual snow syndrome | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: In a double-blind, randomized and placebo-controlled longitudinal experiment, the investigators will use real-time functional magnetic resonance imaging (rtfMRI) neurofeedback to teach patients to downregulate activity in different regions of the visual cortex.
  50 patients (25 in each arm)
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients group 1 (Active Comparator): This group will regulate a brain region by real-time functional magnetic resonance imaging that is centrally involved in the visual snow syndrome
  Interventions: Other: neurofeedback
- Patients group 2 (Placebo Comparator): This group will regulate a brain region by real-time functional magnetic resonance imaging that is not centrally involved in the visual snow syndrome
  Interventions: Other: neurofeedback

INTERVENTIONS:
Other: neurofeedback — (based on real-time functional magnetic resonance signals)

SUMMARY:
Visual snow (VS) is a distressing, life-impacting condition with unrelenting and persistent disturbing visual phenomena. Disease onset is usually around age 20 and is characterized by continuous perception of innumerable flickering dots (like a 'broken television'). The disease is often accompanied by comorbidities such as migraine, tinnitus, depression and anxiety.

Neuronally, VS patients show cerebral hypermetabolism, resulting in altered neuronal excitability, as well as increased grey matter volume in parts of the visual cortex.

For this pilot study, the investigators aim to recruit VS patients. In a double-blind, randomized and placebo-controlled longitudinal experiment, the investigators will use real-time functional magnetic resonance imaging (rtfMRI) neurofeedback to teach patients to downregulate activity in different regions of the visual cortex.

The investigators hypothesize that neurofeedback will allow patients to learn to downregulate their abnormal visual cortex activity. Moreover, the investigators predict that a stronger downregulation of activity from the lingual gyrus will correlate with a more pronounced decrease in VS symptoms.

DETAILED DESCRIPTION:
Currently, there is no pharmacological or non-pharmacological treatment available that significantly reduces the high disease burden produced by VS. Thus, there is an unmet need for an appropriate intervention to treat patients with VS. In this study, the investigators will:

1. Test if rtfMRI-based neurofeedback could serve as therapeutic option for patients with VS.

   Here, the investigators will examine correlations of neurofeedback regulation success with clinical scores 3 after neurofeedback
2. Examine brain function and structure in patients with VS

Primary and secondary endpoint/outcome(s)

* Primary outcome variable: VS symptom severity before and after rtfMRI, using standardized clinical assessment.
* Secondary outcome variables: fMRI and structural MRI, clinical questionnaires (visual function, anxiety, depression, tinnitus, and migraine), parameters from psychophysical data (assessed before and after neurofeedback).
* Linear Mixed model analysis will be performed (using clinical and imaging data) to estimate the impact of rtfMRI on clinical progression and brain function/structure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with VS (≥ 18 to ≤ 60 years), which can read and sign the informed consent form.
* Male and female
* Healthy controls (≥ 18 to ≤ 60 years), which can read and sign the informed consent form.

Exclusion Criteria:

* MR exclusion criteria (patients only): metallic items in the body (i.e. eye splinter, MR incompatible implants), pacemaker, claustrophobia).
* pregnant participants
* participants suffering from a degenerative disorder of the Central Nervous System, such as Stroke, Multiple Sclerosis, Parkinson's Disease, Alzheimer's Disease and Huntington's Disease and with major psychiatric disorders such as schizophrenia, depression, or anxiety disorder requiring pharmacological treatment (psycho-pharmaca).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
symptom severity | Acute after neurofeedback and 3 months after neurofeedback
  Changes in symptom severity before and after real-time fMRI neurofeedback

SECONDARY OUTCOMES:
Magnetic resonance imaging | before and immediately after the neurofeedback sessions
  Assessment of Magnetic resonance imaging parameters related to brain function and structure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The datasets presented in this study are not readily available because due to Swiss law, the researchers must assess whether the use of the data and coded datasets are within the primary scope of the informed consent. Subject level data is only available upon request and after the researchers have reviewed the purpose of the inquiry. Requests to access the datasets should be directed to Dr. Lars Michels, lars.michels@usz.ch.